CLINICAL TRIAL: NCT02687152
Title: Effect of Arginase Inhibition on Microvascular Endothelial Function in Patients With Type 2 Diabetes and Microvascular Dysfunction.
Brief Title: Arginase Inhibition and Microvascular Endothelial Function in Type 2 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, John Pernow, MD, PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Micro Arginase
Record Dates: First submitted 2016-02-09; First posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — N(omega)-hydroxynorarginine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arginase inhibition (Experimental): N-hydroxyl-nor-L-arginine, i.a. 0.1 mg/min for 120 min
  Interventions: Other: N-hydroxy-nor-L-arginine

INTERVENTIONS:
Other: N-hydroxy-nor-L-arginine

SUMMARY:
The present project is designed to test the hypothesis that arginase contributes to microvascular endothelial dysfunction in patients with type 2 diabetes and microvascular complications.

DETAILED DESCRIPTION:
Background

The development of microvascular complications in diabetes is a complex process, in which endothelial dysfunction is of importance. Emerging evidence suggests that arginase is a key mediator of endothelial dysfunction in type 2 diabetes mellitus (T2DM) by reciprocally regulating nitric oxide bioavailability. The aim of this study was to test the hypothesis that arginase activity is increased and that arginase contributes to microvascular endothelial function in patients with T2DM and microvascular dysfunction.

Method

Microvascular endothelium-dependent and -independent vasodilatation are investigated in patients with T2DM (n =12) and healthy age-matched control subjects (n =12) with laser-Doppler flowmetry during iontophoretic application of acetylcholine and sodium nitroprusside, respectively, before and after intra-arterial administration of the arginase inhibitor N-hydroxy-nor-L-arginine (0.1 mg/min) for 120 min.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes mellitus and microvascular dysfunction defined as microalbuminuria > 3.0 mg/mmol or presence of retinopathy.

Exclusion Criteria:

* Myocardial infarction or unstable angina within the last three months,
* Changed dose of any vasodilator drug during the preceding six weeks,
* Ongoing treatment with warfarin
* Concomitant disease that may have interfered with the possibility for the patients to comply with or complete the study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-03; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in cutaneous microvascular endothelial function | 2 hours
  Laser Doppler flow rate

CONTACTS AND LOCATIONS:
Overall Officials: John Pernow, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No